CLINICAL TRIAL: NCT04486404
Title: Personal Protective Equipmente Needs, Perceptions and Acute Stress Among Healthcare Workers Caring for COVID-19 Patients in South America
Brief Title: Needs, Perceptions and Acute Stress of Healtcare Workers Caring for COVID-19 Patients in South America
Status: Completed | Type: Observational
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Universidad Catolica Santiago de Guayaquil (Other); Universidad de Santander (Other); University of Sao Paulo (Other); Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, PhD, Universidad Miguel Hernandez de Elche
Other Study IDs: 08/04/2020
Record Dates: First submitted 2020-07-23; First posted 2020-07-24 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Acute Stress Disorder
Keywords: COVID-19; Healthcare Personnel; Mental Health; Acute stress; Hospitals; Primary care
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Online survery to healtcare personnel and other professionals in the front-line from Col, Bra and Ec.
  Interventions: Other: Online survey
- Group 2: Online survery to healtcare personnel and other professionals in the front-line from Col, Bra, Ch and Ec.
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — Online survey including questions related to PPE availability, perceptions, emotions and EASE scale (Acute Stress Scale).

SUMMARY:
The pressure on care and the demand for critical decision-making generated by the current SARS-CoV-2 (COVID-19) pandemic, together with the situation of extreme social alarm and the adverse conditions in which care work must be promoted at this time, draw an extreme scenario in which action is urgently needed to alleviate emotional overload, acute stress reactions and other affective pathologies or psychosomatic reactions that may eventually lead to post-traumatic stress situations. This eventuality is being observed massively among professionals from different groups and levels of responsibility.

In the case of healthcare personnel, it should be added that the care of non-COVID19 patients (of all pathologies and conditions) is clearly compromised and it is up to the professionals as a whole to make critical decisions and exercise a professional practice that is radically different from what has usually been done, which may require the application of undesirable triage criteria that are difficult for everyone to assume.

Healthcare professionals and other essential personnel for healthcare and social-healthcare work (including personnel from external companies) are being subjected to emotional tensions and extraordinary, high-intensity work demands. Without professionals who feel supported and with moral strength, care will be even more compromised.

The current scenario makes us think of many critical situations that are occurring as a result of the overload experienced. It is essential to act in order to counteract the devastating effect of this health crisis on health professionals and those who support them in their care work.

DETAILED DESCRIPTION:
Coronavirus 2019 disease - of recent appearance - has become a global public health problem due to its rapid spread, since 11 March declared by WHO as a pandemic. It represents a real challenge for health systems, which at first lack information to organize the response to this situation, effective treatments to combat this lethal infection and with health personnel lacking the necessary security in their daily work to minimize the risk of contagion. The COVID-19 pandemic has caused, up to July 21, more than 609,000 deaths worldwide, 28,422 in Spain. The number of professionals suffering from COVID-19 is high. In Spain it accounts for more than 20% of the total number of people infected.

In this way, health professionals have been taking on a notable role without hardly any intention of doing so. Situations of constant uncertainty and emotional distress have posed a risk to patients and to the quality of care, making health professionals the second most affected by SARS-CoV-2 (COVID-19), which also requires special biosecurity and protection measures.

In a global survey, 52% of the 2711 health workers included reported that at least 1 standard PPE piece was out of stock. For example, in the United States, the Food and Drug Administration and the Centers for Disease Control and Prevention have taken several steps to optimize the use of PPE due to its scarcity. Although professionals in Germany consider that they have been well prepared for the pandemic, there are substantial differences in the availability of PPE depending on the health professional and the setting (outpatient or acute care hospitals). In Spain, 54% of primary health care workers reported that they were not adequately trained to use PPE. No similar studies we found in the local context of South American countries.

Although the incidence of the pandemic has expanded differently in different geographical areas of each country, most hospitals and health centres around the world have had to reorganise themselves to prioritise the care of COVID-19 patients, breaking with their usual work dynamics. To this cause of work stress must be added the uncertainty in which decisions have had to be made and the lack of resources both to treat patients adequately and to protect against possible contagion. Reactions of compassionate fatigue, post-traumatic stress, and moral damage have been observed among health professionals, which has depended on the expansion of the pandemic, available means, and individual differences in stress response.

These types of responses and reactions to this crisis are natural and affect all staff and all professional levels, including care support staff (IT, supplies, cleaning, etc.). The opposite would be difficult to explain. However, the key question is not the number of professionals who have been emotionally affected as a result of their care work, a circumstance that is aggravated in this crisis but is inherent to the work they do, but rather how many are unable to recover, how their resilience is evolving or to what extent they are able to cope with a possible new outbreak.

Most studies have analysed the emotional responses in a short period of time (approximately one week) coinciding with a specific stage of the crisis. However, studies on community coping with catastrophic situations have described that the psychological response evolves over time resulting in: impact phase, heroic (intensification of efforts), honeymoon (optimism), disillusionment (fatigue) and restoration (recovery pre-crisis levels). Therefore, it is expected that the effects of the pandemic on the psychological and emotional well-being of health professionals will vary as the pandemic evolves.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals, other professionals working in the front-line of COVID-19.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare personnel in the front line of exposure to suspicious and confirmed cases of COVID-19 and healthcare support personnel (administrative assistants, cleaning or security personnel) of these services and units, such as Emergency and Primary Health Care Services, Internal Medicine, Critical Care and Resuscitation, Intermediate Care and any other area designated for the care of such cases.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Acute Stress | 15 days
  Prevalence of acute stress using the Acute Stress Scale (EASE Scale) among healthcare personnel in the front-line caring for COVID-19 patients.
  Score values range from 0 to 30. 0-9 points, good emotional adjustment; 10-14 points, emotional distress; 15-24 points, medium-high emotional overload; > 25 points, extreme acute stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jose J Mira, PhD, Principal Investigator — Universidad Miguel Hernández de Elche
Locations (5):
- Institute for Clinical Effectiveness and Health Policy, Buenos Aires, Argentina
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Universidad de Santander, Bucaramanga, Santander Department, Colombia
- Universidad Católica de Santiago de Guayaquil, Guayaquil, Guayas, Ecuador
- Universidad Miguel Hernández de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Auxemery Y. Treatment of post-traumatic psychiatric disorders: A continuum of immediate, post-immediate and follow-up care mediated by specific psychotherapeutic principles. Clinical experience in French-speaking countries. Encephale. 2018 Nov;44(5):403-408. doi: 10.1016/j.encep.2018.02.003. Epub 2018 Jun 8. PMID 29887301
- [Background] Chen Q, Liang M, Li Y, Guo J, Fei D, Wang L, He L, Sheng C, Cai Y, Li X, Wang J, Zhang Z. Mental health care for medical staff in China during the COVID-19 outbreak. Lancet Psychiatry. 2020 Apr;7(4):e15-e16. doi: 10.1016/S2215-0366(20)30078-X. Epub 2020 Feb 19. No abstract available. PMID 32085839
- [Background] Everly GS Jr, Mitchell JT. The debriefing "controversy" and crisis intervention: a review of lexical and substantive issues. Int J Emerg Ment Health. 2000 Fall;2(4):211-25. PMID 11217152
- [Background] Kang L, Li Y, Hu S, Chen M, Yang C, Yang BX, Wang Y, Hu J, Lai J, Ma X, Chen J, Guan L, Wang G, Ma H, Liu Z. The mental health of medical workers in Wuhan, China dealing with the 2019 novel coronavirus. Lancet Psychiatry. 2020 Mar;7(3):e14. doi: 10.1016/S2215-0366(20)30047-X. Epub 2020 Feb 5. No abstract available. PMID 32035030
- [Background] Khalid I, Khalid TJ, Qabajah MR, Barnard AG, Qushmaq IA. Healthcare Workers Emotions, Perceived Stressors and Coping Strategies During a MERS-CoV Outbreak. Clin Med Res. 2016 Mar;14(1):7-14. doi: 10.3121/cmr.2016.1303. Epub 2016 Feb 4. PMID 26847480
- [Background] Li W, Yang Y, Liu ZH, Zhao YJ, Zhang Q, Zhang L, Cheung T, Xiang YT. Progression of Mental Health Services during the COVID-19 Outbreak in China. Int J Biol Sci. 2020 Mar 15;16(10):1732-1738. doi: 10.7150/ijbs.45120. eCollection 2020. PMID 32226291
- [Background] Mira JJ, Carrillo I, Guilabert M, Lorenzo S, Perez-Perez P, Silvestre C, Ferrus L; Spanish Second Victim Research Team. The Second Victim Phenomenon After a Clinical Error: The Design and Evaluation of a Website to Reduce Caregivers' Emotional Responses After a Clinical Error. J Med Internet Res. 2017 Jun 8;19(6):e203. doi: 10.2196/jmir.7840. PMID 28596148
- [Background] Mira JJ, Carrillo I, Lorenzo S, Ferrus L, Silvestre C, Perez-Perez P, Olivera G, Iglesias F, Zavala E, Maderuelo-Fernandez JA, Vitaller J, Nuno-Solinis R, Astier P; Research Group on Second and Third Victims. The aftermath of adverse events in Spanish primary care and hospital health professionals. BMC Health Serv Res. 2015 Apr 9;15:151. doi: 10.1186/s12913-015-0790-7. PMID 25886369
- [Background] Mitchell JT. Innovative, precise, and descriptive terms for group crisis support services: a United Nations initiative. Int J Emerg Ment Health. 2007 Fall;9(4):247-52. PMID 18459528
- [Background] Scott SD, Hirschinger LE, Cox KR, McCoig M, Hahn-Cover K, Epperly KM, Phillips EC, Hall LW. Caring for our own: deploying a systemwide second victim rapid response team. Jt Comm J Qual Patient Saf. 2010 May;36(5):233-40. doi: 10.1016/s1553-7250(10)36038-7. PMID 20480757
- [Background] Wu P, Fang Y, Guan Z, Fan B, Kong J, Yao Z, Liu X, Fuller CJ, Susser E, Lu J, Hoven CW. The psychological impact of the SARS epidemic on hospital employees in China: exposure, risk perception, and altruistic acceptance of risk. Can J Psychiatry. 2009 May;54(5):302-11. doi: 10.1177/070674370905400504. PMID 19497162
- [Background] Xiang YT, Yang Y, Li W, Zhang L, Zhang Q, Cheung T, Ng CH. Timely mental health care for the 2019 novel coronavirus outbreak is urgently needed. Lancet Psychiatry. 2020 Mar;7(3):228-229. doi: 10.1016/S2215-0366(20)30046-8. Epub 2020 Feb 4. No abstract available. PMID 32032543
- [Derived] Martin-Delgado J, Poblete R, Serpa P, Mula A, Carrillo I, Fernandez C, Vicente Ripoll MA, Loudet C, Jorro F, Garcia Elorrio E, Guilabert M, Mira JJ. Contributing factors for acute stress in healthcare workers caring for COVID-19 patients in Argentina, Chile, Colombia, and Ecuador. Sci Rep. 2022 May 19;12(1):8496. doi: 10.1038/s41598-022-12626-2. PMID 35589975
- [Derived] Martin-Delgado J, Viteri E, Mula A, Serpa P, Pacheco G, Prada D, Campos de Andrade Lourencao D, Campos Pavan Baptista P, Ramirez G, Mira JJ. Availability of personal protective equipment and diagnostic and treatment facilities for healthcare workers involved in COVID-19 care: A cross-sectional study in Brazil, Colombia, and Ecuador. PLoS One. 2020 Nov 11;15(11):e0242185. doi: 10.1371/journal.pone.0242185. eCollection 2020. PMID 33175877
- See also: Be+ Against COVID Second Victims working group website — https://secondvictimscovid19.umh.es/p/home.html
- See also: EASE Scale pre-print — https://www.researchsquare.com/article/rs-39710/v1